CLINICAL TRIAL: NCT04451876
Title: Social Media Use ,Online Health Information Seeking and Knowledge on Hypertension Among Undergraduate Students of Faculty of Medicine and Health Sciences (FMHS), Universiti Putra Malaysia (UPM)
Brief Title: Social Media Use ,Online Health Information Seeking and Knowledge on Hypertension
Status: Completed | Type: Observational
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Aneesa Abdul Rashid, Medical Lecturer and Family Medicine Specialist, Universiti Putra Malaysia
Other Study IDs: UPM 007
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-11

CONDITIONS: Hypertension; Knowledge, Attitudes, Practice; Social Behavior
Keywords: hypertension; online health information; social media
MeSH Terms: conditions — Hypertension; Behavior; Social Behavior

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The percentage of hypertension among adults aged 18 is relatively high which is about 30% in Malaysia. Uncontrolled hypertension will increase the risk of diseases especially cardiovascular disease. However, adults still lack awareness about the importance of knowledge of hypertension. In between, online health information seeking and the use of social media to gather health information have been quite a norm among students. The wide use of this platform has been proven in various researches and studies.

This study will be conducted among the undergraduate students in FMHS, UPM to look at the various socio-demographic factors associated with their level of knowledge on hypertension. Therefore, this may lead to a need to plan awareness programs on hypertension and to increase the knowledge of hypertension among health science students in the future. A cross-sectional study design will be done for this study. All undergraduate students in FMHS, UPM will be selected through simple random sampling. Online questionnaires will be given via the selected student email platform.

However, there are limitations for this study where we only focus on the students of FMHS, UPM. Hence, the results of this study may be limited to them only. The causal relationship cannot be determined by this study design as well. The purpose of this study is to determine the social media use, online health information seeking practices with knowledge on hypertension among undergraduate students in FMHS, UPM, and its associated factors

DETAILED DESCRIPTION:
BACKGROUND Hypertension is a medical condition that acts as an important public health problem worldwide. It contributes to the disease which is mostly seen in primary health care settings such as cardiovascular disease, stroke, kidney failure, and premature death if it is not diagnosed as soon as possible. The World Health Organization (WHO) significantly mentions that an estimation of 1.13 billion people worldwide from poor countries where the healthcare system is weak have been detected with hypertension. Hypertension also puts an enormous financial pressure towards individuals and medical services via utilizing limited resources . Hypertension is predisposed to multiple factors. Such factors vary from country to country and there is also a disparity between urban and rural areas of the same location.

In Malaysia, 30% of adults above 18 have hypertension. Based on another study, it was proven that adults with uncontrolled hypertensive portrayed a higher risk of CVD mortality when compared to normotensive adults. It was reported that there were 3550 of them all caused hypertensive death and based on that 1027 are caused by cardiovascular disease; 771 are caused by heart-specific diseases and 256 by a cerebrovascular specific disease. However, untreated hypertension was stated to be the high risk of all caused death.

Based on a study by Grad I. et al, global knowledge on hypertension among adults is relatively low which is almost 49.2%. Whereas for medium knowledge on hypertension has 38% and only reported that 13% has higher knowledge on hypertension

. Besides, adults also have insufficient knowledge on epidemiology, method of treatment, and avoidance of hypertension(6).In addition, a good understanding of hypertension has also been linked with enhanced compliance with medications and good control of blood pressure.

According to Loiselle (1995), health information behavior is basically defined as a self-regulatory technique used by patients to coordinate transactions between self-related and health-related settings with the goal of balancing instrumental benefits and informative subjective costs. The students use electronic health knowledge to take some essential health-related decisions and actions. Students reported using the health details gathered more as a guide for lifestyle changes (72.4%) and the rest is dealing with healthcare practitioners online about the change in medication and guide of lifestyle changes.

WHO states that many people, primarily in the developing world, have access to online medical information, engage in online groups, buy well-being goods and services.

From the other side, hospital reports are often linked up by health agencies. The search for online health information has been on the increase and the knowledge gained has diverse influences on the healthcare outcomes of human beings. Based on a study conducted on 4504 respondents about mobile health use and perception among Malaysians in Selangor, only 1 in 5 respondents reported using some health-related application or mobile health device. The analysis of the health details that Malaysia is pursuing is still limited. From the point of view of scientific research, not much study has been done on different problems that occurred in the sense of finding health knowledge.

One of the interventional strategies to the elimination of health inequalities is by utilizing social media as a popular way to get health information. Depending on the concepts of loyalty and mutuality, social media promotes the sharing of life-enhancing services, such as health-related knowledge and social ties. In fact, social media sites are activating feedback systems that result in an enhanced degree of self-efficacy, which is vital in sustaining healthier behaviors and adhering to treatment. It becomes a mixture of direct contact and mainstream media which is personalized and responsive. Social networking media, including Facebook, one of the social media networking platforms, has such connectivity features in their architecture. As of 2004, it has been extremely popular with more than 350 million users around the world.

Non-communicable diseases constitute a worldwide crisis that contributes to more than 36 million (63 %) of all mortality globally. Almost 29 million (80%) of such deaths arise in low-and middle-income nations. Increasing use of social media implies a strategy to achieve scalability or even overcome barriers that often impede public health measures. For example, a smartphone-based home glucose monitoring service has been implemented through which community health professionals have given clinical advice for diabetic patients through smartphones.

The social media use, health information seeking, and knowledge on hypertension in Malaysia are not well studied. It is beneficial to have an overview of the social media use, health information seeking and knowledge on hypertension among the students of Faculty of Medicine and Health Science (FMHS), UPM because they are individuals who will work in a healthcare setting in the near future.

In conclusion, knowledge of hypertension is relatively very important to reduce the prevalence of hypertension and to create more awareness among the public. Ways of getting knowledge and online health information like social media are important as it is becoming a popular form of information. This study will be conducted among the students in FMHS, UPM because of the variety of sociodemographic factors present that will be a platform to see the association between the factors and their level of knowledge on hypertension. Moreover, this may be a good start to plan an awareness program on Hypertension and also initiate programs to increase the knowledge of hypertension among the students.

STUDY OBJECTIVE General Objective To determine the social media use, online health information seeking and knowledge on hypertension among students in FMHS, UPM.

Specific Objective I. To determine the socio-demographic factors (age, gender, race, family income status, undergraduate course and year of study) of students of FMHS, UPM. II. To determine the social media use of students among FMHS, UPM. III. To determine the online health information-seeking behavior on hypertension among students of FMHS, UPM. IV. To determine the level of knowledge on hypertension among students of FMHS, UPM. V. To study the association of socio-demographic factors, social media use and online health information seeking on the knowledge of hypertension.

STUDY INSTRUMENTS Study instruments include a questionnaire adapted from a previously published questionnaire. The questionnaire to assess the social media use and health information seeking was adapted from a study about Health Information Seeking and Social Media Use on the Internet among people with Diabetes. The hypertension knowledge questionnaire was adapted from a tool developed to assess hypertension knowledge among urban patients. This questionnaire is prepared in English and is divided into four parts.

ELIGIBILITY:
Inclusion Criteria:

All undergraduate students in the Faculty of Medicine and Health Science (FMHS), Universiti Putra Malaysia (UPM).

Exclusion Criteria:

1. Students who are on long leave
2. Students who have dropped out of the course.
3. Students who are acutely unwell

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: This study will take place at the Faculty of Medicine and Health Sciences, University Putra Malaysia in Serdang, Malaysia. This faculty is one of the 16 faculties in University Putra Malaysia and it has almost 1370 undergraduate health sciences and medical students. This number of students in each course offered is Doctor of Medicine (509), Biomedical Sciences (214), Environmental and Occupational Health (213), Dietetic (138), Nutrition and Community Health (196), Bachelor of Nursing (100).The duration of the study of each course varies from four to five years.
Sampling Method: Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Knowledge on Hypertension | 1 week
  Questionnaire on knowledge of hypertension. Minimum score= 0, Maximum Score=10, the higher score, the better the hypertension knowledge

SECONDARY OUTCOMES:
Social Media | 1 week
  Questionnaire on social media use (no scores, only asks the types and frequency of social media used)
Online Health Seeking on Hypertension | 1 week
  Questionnaire on Online Health Seeking on Hypertension (no scores, only asks if the participants sought any health information online, on what kind of information)

CONTACTS AND LOCATIONS:
Locations (1):
- Universiti Putra Malaysia, Seri Kembangan, Selangor, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided
Sharing of information of students will be aligned with Universiti's rulings.

REFERENCES:
- [Background] Naing C, Yeoh PN, Wai VN, Win NN, Kuan LP, Aung K. Hypertension in Malaysia: An Analysis of Trends From the National Surveys 1996 to 2011. Medicine (Baltimore). 2016 Jan;95(2):e2417. doi: 10.1097/MD.0000000000002417. PMID 26765422
- [Background] Rani R, Mengi V, Gupta RK, Sharma HK. Hypertension and Its Risk Factors - A Cross Sectional Study in an Urban Population of a North Indian District. Public Health Res. 2015;5(3):67-72.
- [Background] Zhou D, Xi B, Zhao M, Wang L, Veeranki SP. Uncontrolled hypertension increases risk of all-cause and cardiovascular disease mortality in US adults: the NHANES III Linked Mortality Study. Sci Rep. 2018 Jun 20;8(1):9418. doi: 10.1038/s41598-018-27377-2. PMID 29925884
- [Background] Grad I, Mastalerz-Migas A, Kilis-Pstrusinska K. Factors associated with knowledge of hypertension among adolescents: implications for preventive education programs in primary care. BMC Public Health. 2015 May 3;15:463. doi: 10.1186/s12889-015-1773-7. PMID 25935154
- [Background] Almas A, Godil SS, Lalani S, Samani ZA, Khan AH. Good knowledge about hypertension is linked to better control of hypertension; a multicentre cross sectional study in Karachi, Pakistan. BMC Res Notes. 2012 Oct 24;5:579. doi: 10.1186/1756-0500-5-579. PMID 23095492
- [Background] Lambert SD, Loiselle CG. Health information seeking behavior. Qual Health Res. 2007 Oct;17(8):1006-19. doi: 10.1177/1049732307305199. PMID 17928475
- [Background] Osei Asibey B, Agyemang S, Boakye Dankwah A. The Internet Use for Health Information Seeking among Ghanaian University Students: A Cross-Sectional Study. Int J Telemed Appl. 2017;2017:1756473. doi: 10.1155/2017/1756473. Epub 2017 Oct 31. PMID 29225620
- [Background] Nangsangna RD, da-Costa Vroom F. Factors influencing online health information seeking behaviour among patients in Kwahu West Municipal, Nkawkaw, Ghana. Online J Public Health Inform. 2019 Sep 19;11(2):e13. doi: 10.5210/ojphi.v11i2.10141. eCollection 2019. PMID 31632607
- [Background] Lee JY, Wong CP, Lee SWH. m-Health views and perception among Malaysian: findings from a survey among individuals living in Selangor. Mhealth. 2020 Jan 5;6:6. doi: 10.21037/mhealth.2019.09.16. eCollection 2020. PMID 32190617
- [Background] Shaya FT, Chirikov VV, Daniel Mullins C, Shematek J, Howard D, Foster C, Saunders E. Social networks help control hypertension. J Clin Hypertens (Greenwich). 2013 Jan;15(1):34-40. doi: 10.1111/jch.12036. Epub 2012 Nov 26. PMID 23282122
- [Background] Shaw RJ, Johnson CM. Health Information Seeking and Social Media Use on the Internet among People with Diabetes. Online J Public Health Inform. 2011;3(1):ojphi.v3i1.3561. doi: 10.5210/ojphi.v3i1.3561. Epub 2011 Jun 22. PMID 23569602
- See also: information on Hypertension by WHO — https://www.who.int/news-room/fact-sheets/detail/hypertension
- See also: National Health and Mobidity Survey, Malaysia — https://mpaeds.my/national-health-and-morbidity-survey-2019/